CLINICAL TRIAL: NCT03846102
Title: MORphine Use in the Fascia Iliaca Compartment Block With UltraSound
Acronym: MORFICUS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID-19 crisis.
Sponsor: Zuyderland Medisch Centrum (Other)
Collaborators: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL60104.096.16; 2016-004698-42 (EudraCT Number); 16T215 (Other: Medical Ethical Committee Zuyderland)
Record Dates: First submitted 2019-02-07; First posted 2019-02-19 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Humans; Anesthetics, Local; Morphine; Pain Management; Analgesia; Pain; Anesthesia, Local; Fascia; Emergency Medicine; Analgesia, Patient-Controlled; Ultrasonography; Femoral Fracture
Keywords: Fascia Iliaca Compartment Block; Peripheral Nerve Block; Elderly; Hip fracture; Levobupivacaïne; Morphine; Emergency Physician; Emergency department; Ultrasound; Pain score; Numerical Rating scale
MeSH Terms: conditions — Agnosia; Pain; Femoral Fractures; Hip Fractures; Emergencies | interventions — Levobupivacaine; Acetaminophen; Morphine

STUDY DESIGN:
Intervention Model Description: double-blinded randomized placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Syringes with either placebo or levobupivacaïne will be prepared under aseptic conditions and blinded by the hospital pharmacy. A supply of at least six syringe packs will be kept in the emergency department. Each pack will contain three different doses of either levobupivacain or placebo, of which one will be used according to the weight of the patient. When medication is used, the nurse, physician or researcher will inform the pharmacy, so new medication can be prepared. The hospital pharmacy will keep track of randomisation and register the allocation to either treatment or placebo. Allocation will remain blinded until all patients are included and all data is included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levobupivacaïne (Experimental): Fascia Iliaca Compartment Block with Levobupivacaine Hydrochloride (weight based dosage and volume)
  Ideal Body Weight : Levobupivacaïne dose (mg) : Dose/kilogram (mg/kg) : Total volume (ml)
  * [<64 kg : 100 mg : 2.0 mg/kg : 40 ml]
  * [65-74 kg : 125 mg : 1.9 mg/kg : 45 ml]
  * [≥ 75 kg : 150 mg : 2.0 mg/kg : 50 ml]
  Acetaminophen 1 gram (tablets) 4 times daily.
  Patient Controlled Analgesia Pump with morphine 1 milligram per dose.
  Interventions: Drug: Levobupivacaine; Drug: Acetaminophen; Drug: Morphine; Procedure: Fascia Iliaca Compartment Block with Levobupivacaine
- Placebo (Placebo Comparator): Fascia Iliaca Compartment Block with placebo (Sodium Chloride 0.9%), similar volume to experimental arm.
  Ideal Body Weight : Total volume (ml)
  * [<64 kg : 40 ml]
  * [65-74 kg : 45 ml]
  * [≥ 75 kg : 50 ml]
  Acetaminophen 1 gram (tablets) 4 times daily.
  Patient Controlled Analgesia Pump with morphine 1 milligram per dose.
  Interventions: Drug: Placebo; Drug: Acetaminophen; Drug: Morphine; Procedure: Fascia Iliaca Compartment Block with placebo

INTERVENTIONS:
Drug: Levobupivacaine — Levobupivacaïne for injection 7.5 mg/kg diluted with Sodium Chloride 0,9%
  Other Names: Chirocaïne; Levobupivacaine Hydrochloride
  Arms: Levobupivacaïne
Drug: Placebo — Sodium Chloride 0,9% for injection/infusion.
  Other Names: Placebo (for levobupivacaïne)
  Arms: Placebo
Drug: Acetaminophen — Acetaminophen 500 milligram tablet
  Other Names: Paracetamol
Drug: Morphine — Morphine 1 mg/ml solution for infusion.
  Other Names: Morphine hydrochloride
Procedure: Fascia Iliaca Compartment Block with Levobupivacaine — Ultrasound guided Fascia Iliaca Compartment Block with levobupivacaine placed in the emergency department by an emergency physician.
  Other Names: Fascia Iliaca Compartment Block; FIC Block
  Arms: Levobupivacaïne
Procedure: Fascia Iliaca Compartment Block with placebo — Ultrasound guided Fascia Iliaca Compartment Block with placebo placed in the emergency department by an emergency physician.
  Other Names: Fascia Iliaca Compartment Block; FIC Block
  Arms: Placebo

SUMMARY:
Appropriate management of analgesia for proximal femoral fractures is a common problem in the emergency department (ED). Side effects from morphine usage such as nausea, vomiting, respiratory depression, sedation, and obstipation are especially pronounced in elderly. Fascia Iliaca Compartment Block (FICB) holds promise as a simple and safe, and effective alternative method to reduce pain. Local anaesthetic injected in the anatomic space underlying the fascia iliaca, spreads to block the nerves traversing it. This regional anaesthesia includes the femoral nerve. Previous studies in the ED showed promise but lacked blinding, involved low numbers of subjects, or did not use ultrasound localisation of the injection site. The latter is becoming common practice. In this randomised placebo controlled trial the FICB with ultrasound localisation of injection of levobupivacaïne will be compared to the FICB with placebo. It aims to prove that less morphine is used in the intervention group. Other research parameters are pain scores and minor adverse events related to morphine use.

DETAILED DESCRIPTION:
Proximal femoral fractures are common in the ED. A major challenge in such subjects is pain management. Suboptimal pain control is associated with stress, a prolonged hospital stay and delirium. Pain or fear of pain can limit early mobilisation, an important goal in treatment. Therefore early pain management is essential. Standard analgesic care consists of acetaminophen, opiates and/or Non-steroidal anti-inflammatory drugs (NSAID's). Opiates can cause respiratory depression, constipation, drowsiness, nausea and vomiting. Especially elderly patients are at risk for these side effects Regional nerve blocks are increasingly being adopted as an alternative pain management to systemic analgesia in the ED. One of such is the Fascia Iliaca Compartment Block (FICB). This is safe and simple to perform. Results from studies, despite lacking ultrasound guidance are promising. No permanent disability resulted from the few minor complications that have been reported. These include bladder perforation, pneumoretroperitoneum and neuropathy of the femoral nerve. Furthermore no additional treatment was necessary. Ultrasound prevents occurrence of such complications.

The studies that have compared this specific block to standard analgesia have shown that regional anaesthesia may be superior. However these studies have low inclusion numbers and lack of randomisation and/or blinding.. Literature up until now has used the numerical rating scale (NRS) as a primary outcome. Although the NRS is a very trustworthy method of measuring pain, the score is a subjective outcome Morphine consumption on the other hand is more objective.

The FICB involves the anatomic space situated at the level of the groin in which important nerves that supply the hip joint lie. Anteriorly the space is covered by the iliac fascia. It is therefore known as the fascia iliaca compartment. By introducing a large volume of local anaesthetic solutions, the femoral, lateral femoral cutaneous and to a lesser extent the obturator nerve are anesthetized. Solutions can spread easily within the compartment. Therefore a safe position injection site can be chosen, minimizing the risk of intravascular injection and nerve damage. The classic position for injection is about 3 centimetres lateral from the femoral nerve. In the original FICB the injection site is determined by using landmarks. The fascia iliaca compartment is then approached by introducing a blunt needle, which enables the physician to feel a 'pop' twice. The first pop is felt when the fascia lata is pierced, the second when the fascia iliaca is passed.

Most ED's nowadays have access to ultrasound. When used for FICB placement, the local anaesthetic solution is visualized as it is introduced into the space. Therefore a higher chance of successful placement of agent and a lower risk of complications can be expected. So far no large double blind randomised placebo controlled trials have evaluated morphine use in ultrasound guided placement of local anaesthetic agents with FICB in the ED. This study is designed as such. Total morphine use will be taken as the primary outcome, administered in the form of patient controlled analgesia (PCA).

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with a proximal femoral fracture (femoral neck, trochanteric and sub trochanteric femoral fracture) upon arrival at the ED.

Exclusion Criteria:

1. No informed consent patient
2. Skin infection at injection site(s)
3. Morphine allergy
4. Levobupivacaïne allergy
5. Operation within an hour after admission
6. Inability to understand and quantify pain on a NRS
7. History of dementia
8. Neurological deficit of fractured leg upon arrival at the ED
9. Trauma with multiple fractures (more than 1)
10. Risk of compartment syndrome of ipsilateral lower leg
11. Proximal femoral fracture with other definitive treatment than operation
12. Transfer to another hospital
13. Actual morphine use
14. Distracting pain in other location than hip
15. Pregnancy
16. No physician/nurse available for procedure.
17. BMI > 40
18. Saturation < 90%
19. Previously unreported hypotension (systolic blood pressure < 100 mmHg)
20. ASA IV or higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
Mean morphine consumption in milligrams per hour with PCA pump, extracted from PCA-pump memory (mg / hour). | From FICB placement up to 6 hours.
  The primary objective is to assess if ultrasound guided FICB with levobupivacaïne results in reduced morphine consumption in ED patients with a proximal femoral fracture at six hours after FICB placement. The morphine consumption will be extracted from the memory from the PCA pump.

SECONDARY OUTCOMES:
Morphine consumption in milligrams per hour at each hour in the time preceding operation. (mg / hour) | Time from FICB placement until operation, up to 24 hours. Time point: each hour
  To assess if there is a difference in morphine consumption at different time points in the time until operation. Data will be extracted from PCA pump memory.
Average of PCA-pump requests for morphine per hour (presses / hour) | Time from FICB placement until operation, up to 24 hours. Time point: each hour
  The amount of times per hour a patient presses the PCA-pump to receive a bolus of morphine preoperatively.
Average time to first morphine administration with PCA-pump (minutes) | Time from FICB placement until operation, up to 24 hours.
  Average time until patient requests first morphine dose by pressing PCA-pump button.
Average pain score at different time points. | Time from FICB placement until operation, up to 24 hours. Time point: each hour
  Pain scores will be reported with the Numerical Rating Scale (NRS). The NRS is a 11 point scale that is used in the hospital pain protocol. 0 equals to no pain at all, 10 is the worst pain one can imagine. It is regarded as a reliable instrument for pain assessment in patients. Patients will be asked to keep track of their pain score at different time points, starting after FICB placement. They will be asked to report their pain score hourly until 22.00h and from 7.00h the next day. The pain scores will be measured with a dedicated android application, with which patients are asked to self-report their hourly pain scores. When patients are asleep no NRS will be recorded, unless they are awake. Also nurses will report pain scores following their normal rounds when changing shifts. A sleeping patient will be regarded as having a low pain score.
Difference in pain scores at movement. | Time from FICB placement until operation, up to 24 hours. Time point: each hour
  The ED or ward nurse will ask and record the NRS when mobilising patients when necessary. Such situations include for example: bedpan for micturition or stools and bed to bed transfer. The recorded data will include time point, situation and NRS.
  Pain scores will be reported with the Numerical Rating Scale (NRS). The NRS is a 11 point scale that is used in the hospital pain protocol. 0 equals to no pain at all, 10 is the worst pain one can imagine.
Patients with occurence of NRS > 3. | Time from FICB placement until operation, up to 24 hours. Time point at 24 hours.
  The number of patient with a NRS > 3, recorded by the patient in the preoperative time.
Number of patients with a delirium in preoperative period. | Time from FICB placement until operation, up to 24 hours. Time point at 24 hours.
  The Delirium Observation Screening (DOS) scale is a validated screening tool for detecting delirium in hospitalised patients. In this hospital the DOS scale is routinely screened three times daily by ward nurses. The DOS will also be reported for participating patients in the preoperative period. Subjects with a reported DOS of ≥ 3 are regarded as being at high risk for having a delirium.
The number of patients with morphine related side effects. | This will be assessed by the nurse at the rounds each shift up to 3 times daily until operation or up to 24 hours.
  A patient will be regarded of having a side effect of morphine in case of any of the following:
  * Occurrence of nausea
  * Occurrence of vomiting
  * Administration of antiemetic medication
  * Episode of respiratory depression (< 10 breaths/minute)
  * Episode of new hypoxia (SaO2 < 90 % )
  * Administration of naloxone, which will be registered by the nurse on the CRF.
  * Episodes of new hypotension. In this trial hypotension is defined as a systolic blood pressure <90 mmHg, mean arterial pressure <60 mmHg or a drop in systolic blood pressure >40 mmHg.
  * Sedation score > 1. This wil be reported by the nurse with the Pasero Opioïd Induced Sedation Scale, as is prescribed by hospital protocol. S = normal sleep, 1 = drowsy but easy to rouse, 2 = sedated and difficult to rouse, and 3 = unconscious).
Number of patients with treatment-related adverse events as assessed by CTCAE v4.0. | Time from FICB placement until operation, up to 24 hours.
  Adverse events relating to the fascia iliaca compartment block or morphine use will be reported.
Time spent on FICB placement in seconds. | The time from needle entering patient, until procedure is terminated by the emergency physician.
  The duration of ultrasound guided FICB placement will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Sanne Postma, MD, Principal Investigator — Zuyderland Medical Center
Locations (1):
- Zuyderland Medisch Centrum, Heerlen, Zuid Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hughes SG. Prescribing for the elderly patient: why do we need to exercise caution? Br J Clin Pharmacol. 1998 Dec;46(6):531-3. doi: 10.1046/j.1365-2125.1998.00842.x. No abstract available. PMID 9862240
- [Result] Cherny N, Ripamonti C, Pereira J, Davis C, Fallon M, McQuay H, Mercadante S, Pasternak G, Ventafridda V; Expert Working Group of the European Association of Palliative Care Network. Strategies to manage the adverse effects of oral morphine: an evidence-based report. J Clin Oncol. 2001 May 1;19(9):2542-54. doi: 10.1200/JCO.2001.19.9.2542. PMID 11331334
- [Result] Chau DL, Walker V, Pai L, Cho LM. Opiates and elderly: use and side effects. Clin Interv Aging. 2008;3(2):273-8. doi: 10.2147/cia.s1847. PMID 18686750
- [Result] Wheeler M, Oderda GM, Ashburn MA, Lipman AG. Adverse events associated with postoperative opioid analgesia: a systematic review. J Pain. 2002 Jun;3(3):159-80. doi: 10.1054/jpai.2002.123652. No abstract available. PMID 14622770
- [Result] Groot L, Dijksman LM, Simons MP, Zwartsenburg MM, Rebel JR. Single Fascia Iliaca Compartment Block is Safe and Effective for Emergency Pain Relief in Hip-fracture Patients. West J Emerg Med. 2015 Dec;16(7):1188-93. doi: 10.5811/westjem.2015.10.28270. Epub 2015 Dec 14. PMID 26759680
- [Result] Ritcey B, Pageau P, Woo MY, Perry JJ. Regional Nerve Blocks For Hip and Femoral Neck Fractures in the Emergency Department: A Systematic Review. CJEM. 2016 Jan;18(1):37-47. doi: 10.1017/cem.2015.75. Epub 2015 Sep 2. PMID 26330019
- [Result] Kearns R, Macfarlane A, Grant A, Puxty K, Harrison P, Shaw M, Anderson K, Kinsella J. A randomised, controlled, double blind, non-inferiority trial of ultrasound-guided fascia iliaca block vs. spinal morphine for analgesia after primary hip arthroplasty. Anaesthesia. 2016 Dec;71(12):1431-1440. doi: 10.1111/anae.13620. Epub 2016 Oct 7. PMID 27714758
- [Result] Birnbaum A, Schechter C, Tufaro V, Touger R, Gallagher EJ, Bijur P. Efficacy of patient-controlled analgesia for patients with acute abdominal pain in the emergency department: a randomized trial. Acad Emerg Med. 2012 Apr;19(4):370-7. doi: 10.1111/j.1553-2712.2012.01322.x. PMID 22506940
- [Result] Walder B, Schafer M, Henzi I, Tramer MR. Efficacy and safety of patient-controlled opioid analgesia for acute postoperative pain. A quantitative systematic review. Acta Anaesthesiol Scand. 2001 Aug;45(7):795-804. doi: 10.1034/j.1399-6576.2001.045007795.x. PMID 11472277
- [Result] Auroy Y, Benhamou D, Bargues L, Ecoffey C, Falissard B, Mercier FJ, Bouaziz H, Samii K. Major complications of regional anesthesia in France: The SOS Regional Anesthesia Hotline Service. Anesthesiology. 2002 Nov;97(5):1274-80. doi: 10.1097/00000542-200211000-00034. PMID 12411815
- [Result] Blackford D, Westhoffen P. Accidental bladder puncture: a complication of a modified fascia iliaca block. Anaesth Intensive Care. 2009 Jan;37(1):140-1. No abstract available. PMID 19157368
- [Result] Atchabahian A, Brown AR. Postoperative neuropathy following fascia iliaca compartment blockade. Anesthesiology. 2001 Mar;94(3):534-6. doi: 10.1097/00000542-200103000-00029. No abstract available. PMID 11374619
- [Result] Shelley BG, Haldane GJ. Pneumoretroperitoneum as a consequence of fascia iliaca block. Reg Anesth Pain Med. 2006 Nov-Dec;31(6):582-3. doi: 10.1016/j.rapm.2006.08.009. No abstract available. PMID 17138203
- [Result] Barrington MJ, Kluger R. Ultrasound guidance reduces the risk of local anesthetic systemic toxicity following peripheral nerve blockade. Reg Anesth Pain Med. 2013 Jul-Aug;38(4):289-99. doi: 10.1097/AAP.0b013e318292669b. PMID 23788067
- [Result] Morrison RS, Dickman E, Hwang U, Akhtar S, Ferguson T, Huang J, Jeng CL, Nelson BP, Rosenblatt MA, Silverstein JH, Strayer RJ, Torrillo TM, Todd KH. Regional Nerve Blocks Improve Pain and Functional Outcomes in Hip Fracture: A Randomized Controlled Trial. J Am Geriatr Soc. 2016 Dec;64(12):2433-2439. doi: 10.1111/jgs.14386. Epub 2016 Oct 27. PMID 27787895
- [Result] Morrison RS, Magaziner J, Gilbert M, Koval KJ, McLaughlin MA, Orosz G, Strauss E, Siu AL. Relationship between pain and opioid analgesics on the development of delirium following hip fracture. J Gerontol A Biol Sci Med Sci. 2003 Jan;58(1):76-81. doi: 10.1093/gerona/58.1.m76. PMID 12560416
- [Result] Rashid A, Beswick E, Galitzine S, Fitton L. Regional analgesia in the emergency department for hip fractures: survey of current UK practice and its impact on services in a teaching hospital. Emerg Med J. 2014 Nov;31(11):909-13. doi: 10.1136/emermed-2013-202794. Epub 2013 Jul 22. PMID 23878064
- [Result] Dalens B, Vanneuville G, Tanguy A. Comparison of the fascia iliaca compartment block with the 3-in-1 block in children. Anesth Analg. 1989 Dec;69(6):705-13. PMID 2589650
- [Result] Hogh A, Dremstrup L, Jensen SS, Lindholt J. Fascia iliaca compartment block performed by junior registrars as a supplement to pre-operative analgesia for patients with hip fracture. Strategies Trauma Limb Reconstr. 2008 Sep;3(2):65-70. doi: 10.1007/s11751-008-0037-9. Epub 2008 Sep 2. PMID 18762870
- [Result] Revill SI, Robinson JO, Rosen M, Hogg MI. The reliability of a linear analogue for evaluating pain. Anaesthesia. 1976 Nov;31(9):1191-8. doi: 10.1111/j.1365-2044.1976.tb11971.x. PMID 1015603
- [Result] Abrahams MS, Aziz MF, Fu RF, Horn JL. Ultrasound guidance compared with electrical neurostimulation for peripheral nerve block: a systematic review and meta-analysis of randomized controlled trials. Br J Anaesth. 2009 Mar;102(3):408-17. doi: 10.1093/bja/aen384. Epub 2009 Jan 26. PMID 19174373
- [Result] Huang JJ, Taguchi A, Hsu H, Andriole GL Jr, Kurz A. Preoperative oral rofecoxib does not decrease postoperative pain or morphine consumption in patients after radical prostatectomy: a prospective, randomized, double-blinded, placebo-controlled trial. J Clin Anesth. 2001 Mar;13(2):94-7. doi: 10.1016/s0952-8180(01)00219-7. PMID 11331167
- [Result] Mouzopoulos G, Vasiliadis G, Lasanianos N, Nikolaras G, Morakis E, Kaminaris M. Fascia iliaca block prophylaxis for hip fracture patients at risk for delirium: a randomized placebo-controlled study. J Orthop Traumatol. 2009 Sep;10(3):127-33. doi: 10.1007/s10195-009-0062-6. Epub 2009 Aug 19. PMID 19690943
- [Result] Petre BM, Roxbury CR, McCallum JR, Defontes KW 3rd, Belkoff SM, Mears SC. Pain reporting, opiate dosing, and the adverse effects of opiates after hip or knee replacement in patients 60 years old or older. Geriatr Orthop Surg Rehabil. 2012 Mar;3(1):3-7. doi: 10.1177/2151458511432758. PMID 23569691
- [Result] Fletcher AK, Rigby AS, Heyes FL. Three-in-one femoral nerve block as analgesia for fractured neck of femur in the emergency department: a randomized, controlled trial. Ann Emerg Med. 2003 Feb;41(2):227-33. doi: 10.1067/mem.2003.51. PMID 12548273
- [Result] Foss NB, Kristensen BB, Bundgaard M, Bak M, Heiring C, Virkelyst C, Hougaard S, Kehlet H. Fascia iliaca compartment blockade for acute pain control in hip fracture patients: a randomized, placebo-controlled trial. Anesthesiology. 2007 Apr;106(4):773-8. doi: 10.1097/01.anes.0000264764.56544.d2. PMID 17413915
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043
- See also: Guideline anticoagluants and regional anestesia and peripheral nerve blocks of the Dutch Society of Anesthesiology — https://www.anesthesiologie.nl/uploads/files/KD_RL_Neuraxisblokkade.pdf